CLINICAL TRIAL: NCT04869995
Title: Behav'Robot: Understanding the Surgeon Behavior During Robot-assisted Surgery (a Qualitative Study)
Brief Title: Behav'Robot: Understanding the Surgeon Behavior During Robot-assisted Surgery
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Troyes (Other)
Responsible Party: Sponsor
Other Study IDs: BehavRobot
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Robotic Surgical Procedures
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention: Senior abdominal and pelvic cavity surgeons (i.e., visceral surgeons, gynecologist surgeons, and urologists) having completed their robot-assisted surgery training, and commonly doing laparoscopic surgery.
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — An individual semi-structured interview per surgeon, according to an interview guide.

SUMMARY:
Robot-assisted surgery is spreading since the last decade, but little is known about the impact of the use of the robot on surgeon practices and behavior in the operation theatre.

Interviewing senior surgeons trained for doing robot-assisted surgery, this qualitative study is expected to provide new insights to understand the surgeons' behavioral changes when using a robot.

This study will contribute to improving training programs in robot-assisted surgery.

ELIGIBILITY:
Inclusion Criteria:

* Senior abdominal and pelvic cavity surgeons (i.e., visceral surgeons, gynecologist surgeons, or urologists).
* Having completed a robot-assisted training
* Commonly doing laparoscopic surgery

Exclusion Criteria:

* Those who refuse to participate in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study participants will comprise senior abdominal and pelvic cavity surgeons (i.e., visceral surgeons, gynecologist surgeons, and urologists) having completed their robot-assisted surgery training, and commonly doing laparoscopic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Elicitation of the surgeons' perception | = interview duration (about 30 minutes)
  Elicitation of the surgeons' perception of practices and behavior changes when doing robot-assisted surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Troyes, Troyes, Grand Est, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cormi C, Parpex G, Julio C, Ecarnot F, Laplanche D, Vannieuwenhuyse G, Duclos A, Sanchez S. Understanding the surgeon's behaviour during robot-assisted surgery: protocol for the qualitative Behav'Robot study. BMJ Open. 2022 Apr 7;12(4):e056002. doi: 10.1136/bmjopen-2021-056002. PMID 35393313